CLINICAL TRIAL: NCT03574038
Title: Transcranial Electrical Stimulation in Stroke EaRly After Onset Clinical Trial
Brief Title: Transcranial Direct Current Stimulation as a Neuroprotection in Acute Stroke
Acronym: TESSERACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Mersedeh Bahr Hosseini, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-000421
Record Dates: First submitted 2018-05-30; First posted 2018-06-29 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Traditional 3+3 (rule-based, modified Fibonacci) dose escalation design
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Transcranial Direct Current Stimulation (Active Comparator): Transcranial Direct Current Stimulation
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham Stimulation (Sham Comparator): Sham Stimulation
  Interventions: Other: Sham Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Patients will be randomized to active treatment (C-tDCS) vs sham stimulation in a 3:1 ratio. There will be 6 dose tiers, reflecting increasing intensity and duration of stimulation: Tier 1 - 1 mA, single 20 - min cycle; Tier 2- 2 mA, single 20 min cycle; Tier 3 - 1 mA, 2 cycles of 20 min/20 min off; Tier 4- 2 mA, 2 cycles of 20 min/20 min off; Tier 5 - 1 mA, 3 cycles of 20 min/20 min off; Tier 6 - 2 mA, 3 cycles of 20 min/20 min off.
  Other Names: C-tDCS
  Arms: Transcranial Direct Current Stimulation
Other: Sham Stimulation — Patients will be randomized to active treatment (C-tDCS) vs sham stimulation in a 3:1 ratio. Patients in the sham stimulation arm at all the tiers will have the cap and electrodes in place, and sham switch moved but without prolonged delivery of electrical stimulation.
  Arms: Sham Stimulation

SUMMARY:
This proposal is a prospective, single-center, dose-escalation safety, tolerability, feasibility and potential efficacy study of transcranial direct current stimulation (tDCS) in acute stroke patients with substantial salvageable penumbra due to a large vessel occlusion who are ineligible for intravenous thrombolysis and endovascular therapy.

DETAILED DESCRIPTION:
This is a single center, sham-controlled, dose escalation study where cathodal tDCS is delivered to threatened but not yet irreversibly damaged (penumbral) tissue in patients with large vessel occlusion who are not eligible for blood flow restoring recanalization procedures. Patients will be randomized in a 3:1 design, to cathodal versus sham (control) stimulation, at each six designed dose tiers. The dose tiers will be increasing in both intensity and duration of the stimulation.

The occurrence of symptomatic intracranial hemorrhage will determine the pace of the escalation through the dose tiers.

ELIGIBILITY:
Inclusion criteria:

1. New focal neurologic deficit consistent with AIS
2. NIHSS≥4 or NIHSS <4 in the presence of disabling deficits
3. Age>18;
4. Presence of any cortical vessel occlusion including ICA, branches of MCA, Anterior Cerebral artery (ACA), Posterior Cerebral artery (PCA), Posterior-Inferior cerebellar artery (PICA);
5. Presence of salvageable penumbra with Tmax> 6 sec/ ischemic core volume (ADC < 620 μm2/s or rCBF< 30%) ≥ 1.2
6. Patient ineligible for IV tPA, per national AHA/ASA Guidelines
7. Patient ineligible for endovascular therapy per AHA/ASA national Guidelines - one or more of: poor prestroke functional status (mRS score >1), mild neurological symptoms (NIHSS <6), large ischemic core (ASPECTS <6), thrombectomy not technically performable due to severe vessel tortuosity, cervical artery chronic occlusion, or other unfavorable angioarchitectural features that preclude endovascular access to the target intracranial vessel. 8) Subject is able to be treated with tDCS within 24 hours of last known well time;

9) A signed informed consent is obtained from the patient or patient's legally authorized representative

Exclusion criteria

1. Acute intracranial hemorrhage
2. Evidence of a large Ischemic core volume (ADC < 620 μm2/s or rCBF< 30%) ≥ 100
3. Presence of tDCS contraindications - electrically or magnetically activated intracranial metal and non-metal implants.
4. Severe MR contrast allergy or renal dysfunction with eGFR<30ml/min, precluding MRI gadolinium or CT iodine contrast
5. Pregnancy
6. Signs or symptoms of acute myocardial infarction, including EKG findings, on admission
7. Suspicion of aortic dissection on admission
8. History of seizure disorder or new seizures with presentation of current stroke
9. Evidence of any other major life-threatening or serious medical condition that would prevent completion of the study protocol including attendance at the 3-month follow-up visit
10. Concomitant experimental therapy
11. Preexisting scalp lesion at the site of the stimulation or presence of skull defects (may alter current flow pattern)
12. Preexisting coagulopathy, consist of platelet count of ≤ 100, INR ≥ 3, PTT ≥ 90.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mersedeh Bahr Hosseini, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California- Los Angeles (UCLA), Los Angeles, California, United States

REFERENCES:
- [Derived] Bahr-Hosseini M, Nael K, Unal G, Iacoboni M, Liebeskind DS, Bikson M, Saver JL; TESSERACT Trial Group. High-definition Cathodal Direct Current Stimulation for Treatment of Acute Ischemic Stroke: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2319231. doi: 10.1001/jamanetworkopen.2023.19231. PMID 37342040

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The first 4 patients (3 Active and 1 Sham) were assigned to Tier 1 (1mA of C-tDCS for 20 min) of the study, and the next 6 patients (4 Active and 2 Sham) were assigned to Tier 2 (2mA of C-tDCS for 20 min) of the study.
Groups:
- High-definition Cathodal Transcranial Direct Current Stimulation (HD C-tDCS)-Tier 1: The first 4 patients were randomized to 1mA of HD C-tDCS for 20 min vs. sham stimulation in a 3:1 ratio.
  A total of 3 patients received active stimulation.
- High-definition Cathodal Transcranial Direct Current Stimulation (HD C-tDCS)-Tier 2: The next 6 patients were randomized to 2mA of HD C-tDCS for 20 min vs. sham stimulation in a 3:1 ratio. A total of 4 patients received active stimulation.
- Sham Stimulation: Sham Stimulation
  Sham Stimulation: A total of 3 patients were enrolled in the Sham arm at Tier 1 and 2. Patients in sham arm had the cap and electrodes in place but without any delivery of electrical stimulation.
Period: Overall Study
Arm/Group | High-definition Cathodal Transcranial Direct Current Stimulation (HD C-tDCS)-Tier 1 | High-definition Cathodal Transcranial Direct Current Stimulation (HD C-tDCS)-Tier 2 | Sham Stimulation
Started | 3 (Patients) | 4 (Patients) | 3 (Patients)
Completed | 3 (Patients) | 4 (Patients) | 3 (Patients)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- High-definition Cathodal Transcranial Direct Current Stimulation: High-definition Cathodal Transcranial Direct Current Stimulation
- Total: Total of all reporting groups
Arm/Group | High-definition Cathodal Transcranial Direct Current Stimulation | Sham Stimulation | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: Year] | 75 (19.6) | 77 (12) | 75 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 2 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety Outcome: Rate of Symptomatic Intracranial Hemorrhage (SICH) in the Active Treatment Arms Compared to Sham Arm
Description: The presence of SICH will be assessed on 24-hour post-stimulation scan. SICH will be defined as an intracranial parenchymal hemorrhage, subarachnoid hemorrhage, or intraventricular hemorrhage with an increase of 4 or more points on the National Institute of Health Stroke Scale (NIHSS) within 24 hours of stimulation.The treatment will be considered to have exhibited adequate safety if tDCS results in lower or equivalent rates of SICH compared to sham.
  The NIHSS is a validated quantitative assessment tool to measure stroke-related neurological deficits and ranges from 0 (no neurological deficits) to a maximum of 42, indicative of a very severe level of impairment.
Time Frame: At 24-hour post-stimulation
Population: One SICH occurred in a Tir 2 patient due to a rupture of mycotic aneurysm causing subarachnoid hemorrhage. This misenrollment was later deemed to be a protocol deviation due to not meeting the entry criteria.
Measure: Count of Participants; unit: Participants
Groups:
- Active Stimulation-Tier 1: High-definition Cathodal Transcranial Direct Current Stimulation (1mA-20min)
- Active Stimulation-Tier 2: High-definition Cathodal Transcranial Direct Current Stimulation (2mA-20min)
- Sham Stimulation: Sham Stimulation
  Sham Stimulation: 3 patients were enrolled in the Sham arm: Patients had the cap and electrodes in place but without any delivery of electrical stimulation.
Arm/Group | Active Stimulation-Tier 1 | Active Stimulation-Tier 2 | Sham Stimulation
Number analyzed (Participants) | 3 | 4 | 3
Participants | 0 | 1 | 0

2. Primary Outcome: Feasibility Outcome: Speed With Which HD C-tDCS Was Implemented
Description: The median time from enrollment to HD C-tDCS initiation in the last 4 enrolled patients included three Active-Tier 2 patients and one sham.
Time Frame: Time from randomization to tDCS initiation assessed up to 30 minutes
Population: The time from enrollment to HD C-tDCS initiation in the last 4 enrolled patients.
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Active Stimulation and Sham: High-definition Cathodal Transcranial Direct Current Stimulation Tier 2 and Sham
Arm/Group | Active Stimulation and Sham
Number analyzed (Participants) | 4
minutes | 12.5 [9 to 15]

3. Primary Outcome: Tolerability Outcome: Percentage of the Patients Completing the Protocol-assigned Stimulation Treatment
Description: Percentage of the patients completing the protocol-assigned stimulation treatment
Time Frame: After 20 minutes of stimulation period
Population: Rate of patients completing the protocol assigned stimulation
Measure: Count of Participants; unit: Participants
Groups:
- Active Stimulation-Tier 1: High-definition Cathodal Transcranial Direct Current Stimulation 1mA-20 min
- Active Stimulation-Tier 2: High-definition Cathodal Transcranial Direct Current Stimulation 2mA-20 min
Arm/Group | Active Stimulation-Tier 1 | Active Stimulation-Tier 2 | Sham Stimulation
Number analyzed (Participants) | 3 | 4 | 3
Participants | 3 | 4 | 3

4. Secondary Outcome: Secondary Safety Outcome: Rate of Early Neurologic Deterioration in All Active Patients Compared to Sham Arm
Description: Early neurological deterioration will be defined as worsening ≥ 4 on NIHSS during the 24-hour period after stimulation without intracranial hemorrhage.
Time Frame: During the 24-hour post-stimulation
Measure: Count of Participants; unit: Participants
Groups:
- Active Stimulation (Tier 1 and 2): High-definition Cathodal Transcranial Direct Current Stimulation
  Transcranial Direct Current Stimulation: Patients were randomized to active treatment (HD C-tDCS) vs sham stimulation in a 3:1 ratio. Seven patients were enrolled in the Active arms: Tier 1 - 1 mA (3 patients), single 20 - min cycle and Tier 2- 2 mA, single 20 min cycle (4 patients).
Arm/Group | Active Stimulation (Tier 1 and 2) | Sham Stimulation
Number analyzed (Participants) | 7 | 3
Participants | 1 | 0

5. Secondary Outcome: Secondary Safety Outcome: Rate of Mortality in All Active Patients Compared to Sham Arm,
Description: Mortality will be defined as death or modified Rankin Scale of 6.
Time Frame: By day 90 post stimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Active Stimulation (Tier 1 and 2) | Sham Stimulation
Number analyzed (Participants) | 7 | 3
Participants | 2 | 1

6. Secondary Outcome: Secondary Safety Outcome: Rate of All Serious Adverse Events Occured During the 90 Days of Study Participation in All Active Patients Compared to Sham.
Description: A serious adverse event is any adverse event that is fatal, is life-threatening, is permanently or substantially disabling, requires or prolongs hospitalization, or requires medical or surgical intervention to prevent one of the above outcomes. The rate of serious adverse events will be compared between the active treatment and sham patients.
Time Frame: By day 90 post-stimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Active Stimulation (Tier 1 and 2) | Sham Stimulation
Number analyzed (Participants) | 7 | 3
Participants | 3 | 2

7. Other Pre Specified Outcome: Per-protocol Exploratory Imaging Efficacy Outcome of Imaging Biomarkers of Neuroprotection and Collateral Enhancement Excluding One Patient With no Penumbra at Baseline on Imaging Core Review and One Patient With Septic Embolization as Stroke Cause.
Description: By comparing the baseline MR/CT imaging with the MR/CT imaging at 2-hour (early) and 24-hour (final) post-stimulation, the following were measured: 1) Final penumbra salvage proportion, 2) Final hypoperfusion lesion reduction, 3) Early relative quantitative cerebral blood volume (qrCBV) enhancement.
Time Frame: At 2-hour and 24-hour post-stimulation
Measure: Median (Inter-Quartile Range); unit: percentage change from baseline
Groups:
- Transcranial Direct Current Stimulation: High-definition Cathodal Transcranial Direct Current Stimulation
  Transcranial Direct Current Stimulation: Patients were randomized to active treatment (HD C-tDCS) vs sham stimulation in a 3:1 ratio. Seven patients were enrolled in the Active arms: Tier 1 - 1 mA (3 patients), single 20 - min cycle and Tier 2- 2 mA, single 20 min cycle (4 patients).
Arm/Group | Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 5 | 3
percentage change from baseline
  Final penumbra salvage proportion percentage | 66 [29 to 80.5] | 0 [0 to 0]
  Final hypoperfusion lesion proportion percentage change | -100 [-100 to -46] | 325 [112 to 412]
  Early qrCBV percentage change | 64 [40 to 110] | -4 [-7 to 1]

8. Other Pre Specified Outcome: Per-protocol Exploratory Clinical Efficacy Outcome: Rate of Functional Independence at 3-month in Active vs. Sham Excluding Two Patients, One With no Penumbra Was Present at Baseline on Imaging Core Review and One With Septic Embolization as Stroke Cause.
Description: Rate of modified Rankin Scale (mRS) of 0-2
Time Frame: At day 90 post stimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Active Stimulation (Tier 1 and 2) | Sham Stimulation
Number analyzed (Participants) | 5 | 3
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: Three months following the study enrollment
Groups:
- Active Stimulation-Tier 1: High-definition Cathodal Transcranial Direct Current Stimulation 1mA-20min
- Active Stimulation-Tier 2: High-definition Cathodal Transcranial Direct Current Stimulation 2mA-20min
- Sham Stimulation: Sham Stimulation
  Patients in sham arm had the cap and electrodes in place but without any delivery of electrical stimulation.
Arm/Group | Active Stimulation-Tier 1 | Active Stimulation-Tier 2 | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/3 | 2/4 | 1/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/4 | 2/3
Other Adverse Events (participants affected / at risk) | 1/3 | 0/4 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Stimulation-Tier 1 (N=3) | Active Stimulation-Tier 2 (N=4) | Sham Stimulation (N=3)
Anticipated serious adverse events (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) — Anticipated serious adverse events were defined as SAEs that are expected and related to acute ischemic stroke complications such as headache, stroke recurrence, pneumonia, systemic blood clots, etc.
Unanticipated serious adverse event (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) — An unanticipated serious adverse event is an SAE that is not deemed an ischemic stroke complication and adjudicated as possibly related to study treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Stimulation-Tier 1 (N=3) | Active Stimulation-Tier 2 (N=4) | Sham Stimulation (N=3)
Anticipated AE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Anticipated adverse events were defined as AEs that are commonly reported and anticipated with tDCS application, such as minor tingling, itchiness, scalp redness, and burning sensation
Unanticipated adverse event (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) — An unanticipated adverse event is an AE that is not commonly reported with tDCS application

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT03574038/Prot_SAP_002.pdf
  • Informed Consent Form (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT03574038/ICF_001.pdf